CLINICAL TRIAL: NCT06345482
Title: A Phase I/II Study of MHB039A for Advanced Solid Tumor to Evaluate the Efficacy and Safety
Brief Title: A Study of MHB039A for Advanced Solid Tumor
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Minghui Pharmaceutical (Hangzhou) Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MHB039A-A-101
Record Dates: First submitted 2024-03-18; First posted 2024-04-03 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MHB039A (Experimental): MHB039A IV every 2 weeks or every 3 weeks (including 5mg/kg、10mg/kg、20mg/kg and 30mg/kg)
  Interventions: Drug: MHB039A

INTERVENTIONS:
Drug: MHB039A — a bispecific antibody

SUMMARY:
Phase I/II open label, multicenter study to evaluate the efficacy and safety of MHB039A in advanced malignant tumors.

DETAILED DESCRIPTION:
This first-in-human, dose escalation and dose expansion study is to evaluate the safety, tolerability, pharmacokinetics (PK), immunogenicity, pharmacodynamics (PD) and anti-tumor activity of MHB039A in patients with advanced solid tumor. The Phase I stage （dose escalation）is to determine the maximum tolerated dose (MTD). The phase II stage （dose expansion）is to determine the recommended Phase 2 dose (RP2D) according to safety and efficacy in specific tumor types.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically documented advanced or metastatic solid tumor that is refractory/relapsed to standard therapies, or for which no effective standard therapy is available, or the subject refuses standard therapy.
* Written and signed informed consent
* Aged 18 years or older
* Eastern Cooperative Oncology Group (ECOG) Performance Score of 0 or 1
* Life expectancy >=3 months

Exclusion Criteria:

* Prior malignancy active within the previous 5 years except for the tumor for which a subject is enrolled in the study, and locally curable cancers that have been apparently cured, (e.g. basal cell skin cancer, or carcinoma in situ of the cervix or others)
* Receiving any chemotherapy within 3 weeks prior to the first dose；or other systemic anticancer therapy within 4 weeks prior to the first dose
* Receiving prior anti-PD-1, anti-PD-L1, anti-CTLA(cytotoxic T-lymphocyte-associated protein)-4 or any other immunotherapy or immune-oncology (IO) agent within 28 days of first dose with MHB039A or experienced a toxicity that led to permanent discontinuation of prior immunotherapy
* Unresolved toxicities from prior anticancer therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Estimated)
Dates: Start 2024-04-16 (Actual); Primary Completion 2028-04-01 (Estimated); Study Completion 2029-06-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of participants with adverse events (AE) | Until 30 days after last dose of MHB039A
  An AE is defined as any untoward medical occurrence in a participant administered a pharmaceutical product temporally associated with the use of study treatment, whether or not considered related to the study treatment.
Number of participants with dose-limiting toxicity (DLT) | At the end of Cycle 1 (each cycle is 21 days for every three weeks cohort and 28 days for every two weeks cohort)
  DLTs will be assessed during the dose-escalation phase and are defined as toxicities related to MHB039A which meet pre-defined severity criteria and occurs within the first cycle of treatment.

SECONDARY OUTCOMES:
Maximum Plasma Concentration (Cmax) of MHB039A | Until 30 days after last dose of MHB039A
  to analysis the serum concentrations of MHB039A at different timepoints to determine the Cmax of MHB039A
The area under the plasma concentration-time curve (AUC) of MHB039A | Until 30 days after last dose of MHB039A
  to analysis the serum concentrations of MHB039A at different timepoints to determine the AUC of MHB039A
To detectable anti-drug antibodies with treated subjects | Until 30 days after last dose of MHB039A
  The immunogenicity of MHB039A will be assessed by the number of subjects who produce anti-drug antibodies (ADAs).
Objective response rate (ORR) | Until 30 days after last dose of MHB039A
  The ORR is defined as the proportion of subjects with confirmed complete remission (CR) or confirmed partial response (PR), based on RECIST Version 1.1.

CONTACTS AND LOCATIONS:
Overall Officials: Shun Lu, MD, Principal Investigator — Shanghai Chest Hospital
Locations (1):
- Shanghai Chest Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No